CLINICAL TRIAL: NCT00076115
Title: Research on the Effectiveness of Risperidone in Bipolar Disorder in Adolescents and Children (REACH): A Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy and Safety of Risperidone for the Treatment of Acute Mania in Bipolar I Disorder
Brief Title: Study to Determine the Effectiveness of Risperidone in Bipolar Disorder in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003631
Record Dates: First submitted 2004-01-14; First posted 2004-01-16 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Bipolar Disorder
Keywords: Bipolar; Mania; Manic; Depressive; Manic Depressive; Bipolar mania; risperidone; adolescents; children
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
A clinical study to determine the safety and effectiveness of risperidone compared with placebo in the treatment of bipolar disorder (manic or mixed type) in children and adolescents aged 10 to 17 years.

DETAILED DESCRIPTION:
Subjects will be aged 10 to 17 years with a diagnosis of Bipolar I disorder and suffering from a current mixed or manic episode. On enrollment, subjects will be assigned to receive 1 of 3 treatments (oral placebo tablets, oral risperidone tablets 0.5 to 2.5 mg, or oral risperidone tablets 3 to 6 mg), which will be administered daily for 3 weeks. Study medication will be increased to the target dosage during the first 7 days, then further increased within the target dosage range reached until maximum tolerated dose is reached by day 10. The maximum tolerated dose will be given for the last 12 days of the study. Risperidone (0.5 to 2.5 mg or 3 to 6 mg doses) or placebo given orally as 0.25, 0.5, 1, 2, 3, or 4 mg tablets (or matching placebo) each day for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Current primary diagnosis of bipolar I disorder, mania or mixed type
* Aged between 10 and 17 years
* Young Mania Rating Scale score greater than or equal to 20 at screening and baseline

Exclusion Criteria:

* Known or suspected history of substance dependence
* Significant risk for suicidal or violent behavior
* Received electroconvulsive treatment within 4 weeks of baseline
* Received a depot antipsychotic within 2 treatment cycle before baseline
* Is unable to swallow medication taken in the form of tablets
* Has a positive result for a urine drug screen done at baseline
* Known or suspected seizure disorder
* Hypothyroidism or hyperthyroidism, unless stabilized on appropriate medication for at least 3 months before screening
* Known or suspected history of hypersensitivity or intolerance to risperidone
* History of a poor antimanic response to risperidone when used in adequate doses for an adequate period as the sole antimanic agent

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2003-12; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The change in the total YMRS score from baseline at the 3-week endpoint

SECONDARY OUTCOMES:
Effects on secondary efficacy variables (YMRS response and onset of maintained response, Clinical Global Impression Scale - Bipolar Disorder [CGI-BP]), safety, tolerability, and pharmacokinetics.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Study to Determine the Effectivness of Risperidone in Bipolar Disorder in Children and Adolescents — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=532&filename=CR003631_CSR.pdf